CLINICAL TRIAL: NCT03904693
Title: Prospective, Multi-center, Double-blind, Randomized, Active-controlled, Triple-dummy, Parallel-group, Group-sequential, Adaptive Phase 3 Clinical Study to Compare the Efficacy and Safety of Macitentan and Tadalafil Monotherapies With the Corresponding Fixed Dose Combination in Subjects With Pulmonary Arterial Hypertension (PAH), Followed by an Open-label Treatment Period With Macitentan and Tadalafil Fixed Dose Combination Therapy
Brief Title: Clinical Study to Compare the Efficacy and Safety of Macitentan and Tadalafil Monotherapies With the Corresponding Fixed-dose Combination Therapy in Subjects With Pulmonary Arterial Hypertension (PAH)
Acronym: A DUE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-077A301; 2014-004786-25 (EudraCT Number); AC-077A301 (Other: Actelion Pharmaceuticals Ltd)
Record Dates: First submitted 2019-04-04; First posted 2019-04-05 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Arterial Hypertension (PAH) (WHO Group 1 PH)
Keywords: Pulmonary Arterial Hypertension; PAH; macitentan; tadalafil; fixed dose combination therapy
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Tadalafil; macitentan

STUDY DESIGN:
Intervention Model Description: In total, approximately 170 subjects are planned to be randomized into study to receive either FDC macitentan/tadalafil or macitentan 10 mg or tadalafil 40 mg given once daily and will also receive matching placebos for two other study treatments. Treatment allocation will be stratified based on prior PAH therapy (i.e., treatment-naïve or treated by an Endothelin receptor antagonist or a Phosphodiesterase type-5 inhibitor as a monotherapy) at baseline. Sample size will be re-estimated at interim analysis if study is not terminated early for efficacy/futility up to sample size of 150-250. After completion of double-blind treatment period, subjects will continue study in an open-label treatment (OLT) period for 24 months, which may be prolonged beyond 24 months until macitentan and tadalafil are accessible at required doses, through other options according to local regulations. All assessments at end of double-blind treatment must be completed before subject enters OLT period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- FDC therapy + Placebo macitentan + Placebo tadalafil (Experimental): Subjects to receive FDC macitentan/tadalafil (macitentan 10 mg and tadalafil 40 mg) plus matching placebos for the two other study treatments.
  Interventions: Drug: FDC macitentan/tadalafil; Drug: Placebo macitentan; Drug: Placebo tadalafil
- Macitentan mono-therapy + Placebo tadalafil + Placebo FDC (Active Comparator): Subjects to receive macitentan 10 mg plus matching placebos for the two other study treatments.
  Interventions: Drug: Macitentan 10 mg; Drug: Placebo FDC; Drug: Placebo tadalafil
- Tadalafil mono-therapy + Placebo macitentan + Placebo FDC (Active Comparator): Subjects to receive tadalafil 40 mg (2 x 20 mg) plus matching placebos for the two other study treatments.
  Interventions: Drug: Tadalafil 40 mg; Drug: Placebo FDC; Drug: Placebo macitentan

INTERVENTIONS:
Drug: FDC macitentan/tadalafil — Film-coated tablet with 10 mg macitentan and 40 mg tadalafil, to be administered orally once daily.
  Other Names: ACT-064992D
  Arms: FDC therapy + Placebo macitentan + Placebo tadalafil
Drug: Macitentan 10 mg — Film-coated tablet with 10 mg macitentan, to be administered orally once daily.
  Other Names: ACT-064992
  Arms: Macitentan mono-therapy + Placebo tadalafil + Placebo FDC
Drug: Tadalafil 40 mg — Film-coated tablet with 40 mg tadalafil (2 x 20 mg tablets), to be administered orally once daily.
  Arms: Tadalafil mono-therapy + Placebo macitentan + Placebo FDC
Drug: Placebo FDC — Matching placebo not containing any active substance but otherwise identical in appearance to the respective active drug tablet, to be administered orally once daily.
  Arms: Macitentan mono-therapy + Placebo tadalafil + Placebo FDC; Tadalafil mono-therapy + Placebo macitentan + Placebo FDC
Drug: Placebo macitentan — Matching placebo not containing any active substance but otherwise identical in appearance to the respective active drug tablet, to be administered orally once daily.
  Arms: FDC therapy + Placebo macitentan + Placebo tadalafil; Tadalafil mono-therapy + Placebo macitentan + Placebo FDC
Drug: Placebo tadalafil — Matching placebo not containing any active substance but otherwise identical in appearance to the respective active drug tablet, to be administered orally once daily.
  Arms: FDC therapy + Placebo macitentan + Placebo tadalafil; Macitentan mono-therapy + Placebo tadalafil + Placebo FDC

SUMMARY:
Combination therapy in pulmonary arterial hypertension (PAH) has been the subject of active investigation for more than a decade, with the benefit of targeting different pathways known to be involved in the pathogenesis of the disease. Adherence to prescribed therapy has an impact on clinical outcomes. Reducing the pill/tablet count and frequency has a major impact on patients' adherence to therapies and therefore the observed clinical outcomes. One way to simplify treatment is to use fixed-dose combination (FDC) products that combine multiple treatments targeting different pathways into a single tablet.

This study aims to demonstrate that the FDC of macitentan and tadalafil is more effective than therapy with 10 mg of macitentan alone or 40 mg of tadalafil alone. This phase 3 study will evaluate the efficacy and safety at 16 weeks of an FDC (macitentan 10 mg and tadalafil 40 mg) against these two PAH-approved therapies given as monotherapy to further confirm the added value of the FDC.

DETAILED DESCRIPTION:
PAH is characterized by a progressive increase in pulmonary arterial pressure (PAP) and in pulmonary vascular resistance (PVR) potentially leading to right heart failure and death. Current PAH-specific therapeutic options include treatments that target the three pathways (endothelin, nitric oxide, and prostacyclin pathways). While combination treatment is common, FDC pills or tablets that combine two or more PAH-specific therapies are not available, thereby requiring participants to take multiple pills/tablets daily. An FDC is an attractive option for PAH participants because it simplifies the treatment regimen by combining two therapies (which would otherwise involve a total of three tablets: one macitentan 10 mg tablet and two tadalafil 20 mg tablets) into a single tablet. Macitentan is an orally active, non-peptide, potent dual endothelin receptor A and B antagonist. Tadalafil is a selective inhibitor of phosphodiesterase type-5 (PDE-5), the enzyme responsible for the degradation of cyclic guanosine monophosphate (cGMP). This study comprises the following consecutive periods: Screening period (lasts up to 30 days), Double-blind treatment period (consists of the titration phase [the first 2 weeks] and the maintenance phase [Week 3 through Week 16]), Open-label treatment period, End-of-Treatment (EOT), Safety follow-up (S-FU) period, and End of Study (EOS). The total study duration for a participant will be up to 30 months. Study assessments like physical examinations, vital signs, right heart catheterization, 6-minute walk test will be performed. Safety will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form (ICF)
* Confirmed diagnosis of symptomatic PAH in WHO FC II or III
* Symptomatic PAH belonging to one of the following subgroups of WHO Group 1 pulmonary hypertension:

  * Idiopathic
  * Heritable
  * Drug- or toxin-induced
  * Associated with connective tissue disease, HIV infection, portal hypertension or congenital heart disease with simple systemic-to-pulmonary shunt with persistent pulmonary hypertension documented by a right heart catheterization (RHC) ≥ 1 year after surgical repair
* PAH diagnosis confirmed by hemodynamic evaluation at rest (through central reading), evaluated within 5 weeks prior to randomization:

  * Mean pulmonary artery pressure (mPAP) ≥ 25 mmHg, AND
  * Pulmonary artery wedge pressure (PAWP) or left ventricular end diastolic pressure (LVEDP) ≤ 15 mmHg, AND
  * Pulmonary vascular resistance (PVR) ≥ 3 WU (i.e., ≥ 240 dyn∙sec∙cm-5)
* Negative vasoreactivity test in idiopathic, heritable, and drug/toxin-induced PAH. (Participants for whom no vasoreactivity test was performed at diagnosis can be eligible if currently treated with PAH therapy for more than 3 months and PAH diagnosis confirmed by hemodynamic evaluation at least 3 months after introduction of their PAH therapy).
* Currently receiving a stable dose of ERA or PDE-5i monotherapy for at least 3 months prior to baseline RHC, within the prespecified doses in the study protocol or no history of PAH-specific treatment
* Participant able to perform the 6MWT with a minimum distance of 100 m and maximum distance of 450 m at Screening
* A woman of childbearing potential must:

  * have negative serum pregnancy test at Screening and a negative urine pregnancy test at Randomization
  * agree to undertake monthly urine pregnancy tests during the study and up to at least 30 days after study treatment discontinuation
  * agree to follow the contraception scheme from Screening up to at least 30 days after study treatment discontinuation

Exclusion Criteria:

* Treatment with a soluble guanylate cyclase stimulator, L-arginine, any form of prostanoids or prostacyclin-receptor agonists (including oral, inhaled, or infused routes) in the 3-month period prior to start of treatment
* Treatment with combination therapy of ERA and PDE-5i in the 3-month period prior to start of treatment or history of intolerance to ERA and PDE-5i combination therapy
* Hypersensitivity to any of the study treatments or any excipient of their formulations
* Treatment with a strong cytochrome P450 3A4 (CYP3A4) inducer in the 1-month period prior to start of treatment
* Treatment with a strong CYP3A4 inhibitor or a moderate dual CYP3A4/CYP2C9 inhibitor or co-administration of a combination of moderate CYP3A4 and moderate CYP2C9 inhibitors in the 1-month period prior to start of treatment
* Treatment with doxazosin
* Treatment with any form of organic nitrate, either regularly or intermittently
* Diuretic treatment initiated or dose changed within 1 week prior to the RHC or start of treatment
* Treatment with another investigational drug in the 3-month period prior to start of treatment
* Body mass index (BMI) > 40 kg/m2 at Screening
* Known presence of three or more of the following risk factors for heart failure with preserved ejection fraction at Screening:

  * BMI > 30 kg/m2
  * Diabetes mellitus of any type
  * Essential hypertension (even if well controlled)
  * Coronary artery disease, i.e. history of stable angina or known more than 50% stenosis in a coronary artery or history of myocardial infarction or history of or planned coronary artery bypass grafting and/or coronary artery stenting
* Known presence of moderate or severe obstructive lung disease any time prior to Screening as specified in study protocol
* Known presence of moderate or severe restrictive lung disease any time prior to Screening as specified in study protocol
* Clinically significant aortic or mitral valve disease; pericardial constriction; restrictive or congestive left-sided cardiomyopathy; life-threatening cardiac arrhythmias; significant left ventricular dysfunction; or left ventricular outflow obstruction, in the opinion of the investigator
* Known permanent atrial fibrillation, in the opinion of the investigator
* Known or suspected uncontrolled thyroid disease (hypo- or hyperthyroidism)
* Documented pulmonary veno-occlusive disease
* Hemoglobin < 100 g/L (<10 g/dL) at Screening
* Known severe hepatic impairment as specified in study protocol
* Serum aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 1.5 × upper limit of normal (ULN) at Screening
* Severe renal impairment at Screening as specified in study protocol
* Systemic hypotension at Screening or Randomization and systemic hypertension at Screening as specified in study protocol
* Acute myocardial infarction or cerebrovascular event (e.g., stroke) within the last 26 weeks prior to Screening
* Known bleeding disorder, in the opinion of the investigator
* Loss of vision in one or both eyes because of non-arteritic anterior ischemic optic neuropathy
* Hereditary degenerative retinal disorders, including retinitis pigmentosa
* History of priapism, conditions that predispose to priapism (example, sickle cell anemia, multiple myeloma, or leukemia) or anatomical deformation of the penis (example, angulation, cavernosal fibrosis, or Peyronie's disease)
* Difficulty swallowing large pills/tablets that would interfere with the ability to comply with study treatment regimen
* Any planned surgical intervention (including organ transplant) during the double-blind treatment period, except minor interventions
* Exercise training program for cardiopulmonary rehabilitation in the 12-week period prior to start of treatment, or planned to be started during the double-blind period of the study
* Pregnant, planning to become pregnant or lactating
* Any known factor or disease that might interfere with treatment adherence, full participation in the study or interpretation of the results as judged by the investigator (e.g., drug or alcohol dependence etc.)
* Known concomitant life-threatening disease with a life expectancy less than (<) 12 months
* Calcium channel blocker treatment initiated, or dose changed within 3 months prior to right heart catheterization (RHC) at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2024-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hany Rofael, MD, Study Director — Janssen, LP
Locations (148):
- United States (26):
  - Providence Medical Foundation, Fullerton, California
  - University of Southern California, Los Angeles, California
  - Piedmont Healthcare, Atlanta, Georgia
  - WellStar Health System, Marietta, Georgia
  - OSF HealthCare Cardiovascular Institute, Peoria, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Norton Healthcare, Louisville, Kentucky
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Washington University School Of Medicine, St Louis, Missouri
  - VA Sierra Nevada Health Care System, Reno, Nevada
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Pitt County Memorial Hospital d/b/a Vidant Medical Center, Greenville, North Carolina
  - Sanford Health, Fargo, North Dakota
  - University of Cincinnati, Cincinnati, Ohio
  - St. Elizabeth Hospital Mercy Bon Secors, Youngstown, Ohio
  - Legacy Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Sanford Health, Sioux Falls, South Dakota
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor Scott White - Plano, Plano, Texas
  - WVU Health Sciences Center, Morgantown, West Virginia
  - University of Wisconsin At Madison, Madison, Wisconsin
  - Medical College of Wisconsin Froedtert Hospital, Milwaukee, Wisconsin
- Australia (3):
  - Royal Adelaide Hospital, Adelaide
  - Pulmonary Arterial Hypertension Clinic, Hobart
  - Core Research Group, Milton
- Brazil (10):
  - Universidade Federal De Minas Gerais - Hospital das Clínicas, Belo Horizonte
  - Instituto das Pequenas Missionárias de Maria Imaculada - Hospital Madre Teresa, Belo Horizonte
  - Fundacao para o Desenvolvimento Medico Hospitalar (UNESP Botucatu), Botucatu
  - Secretaria da Saude do Estado do Ceara - Hospital Doutor Carlos Alberto Studart Gomes, Fortaleza
  - Universidade Federal de Goias - Hospital das Clinicas da UFG, Goiânia
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da PUCRS, Porto Alegre
  - SPDM - Associacao Paulista para o Desenvolvimento da Medicina - Hospital Sao Paulo, São Paulo
  - Hospital Das Clinicas Da Faculdade De Medicina Da USP, São Paulo
- Bulgaria (2):
  - National Heart Hospital, Sofia
  - University Multiprofile Hospital for Active Treatment- UMHAT Sveta Anna AD, Sofia
- Canada (4):
  - Alberta Health Services, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - London Health Sciences Centre, London, Ontario
- China (8):
  - Beijing Anzhen Hospital, Beijing
  - The Second Xiangya Hospital of Central South Hospital, Changsha
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Jiangsu Province Hospital, Nanjing
  - Shanghai Pulmonary Hospital, Shanghai
  - The General Hospital of Northern Theater Command, Shenyang
  - Tianjin Medical University General Hospital, Tianjin
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an
- General University Hospital II.department of Internal Medicine-cardiology and angiology, Prague, Czechia
- Germany (9):
  - Universitatsklinikum Bonn, Bonn
  - Universitatsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitaetsklinikum Giessen, Giessen
  - Universitat Greifswald, Greifswald
  - Universitaetsklinikum Hamburg Eppendorf, Hamburg
  - Thoraxklinik am Universitatsklinikum Heidelberg, Heidelberg
  - Kardiologische Praxis Papenburg, Papenburg
  - Universitaetsklinikum Regensburg, Regensburg
  - Klinikum Würzburg Mitte gGmbH Standort Missioklinik, Würzburg
- Hungary (4):
  - Semmelweis Egyetem,Pulmonológiai Klinika, Budapest
  - Gottsegen György Országos Kardiológiai Intézet, Felnőtt kardiológiai osztály, Budapest
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
  - Szegedi Tudomanyegyetem, Szeged
- Italy (7):
  - Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari, Bari
  - Cardiologia c/o Spedali Civili, Brescia
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera San Gerardo, Monza
  - Ospedale San Francesco, Nuoro
  - IRCCS Policlinico San Matteo, Università degli studi di Pavi, Pavia
  - Policlinico Umberto I, Roma
- Japan (26):
  - The University of Tokyo Hospital, Bunkyō City
  - Chiba University Hospital, Chiba
  - Kyushu University Hospital, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Gunma University Hospital, Gunma
  - Kure Kyosai Hospital, Hiroshima
  - Tokai University Hospital, Isehara
  - Kagoshima University Hospital, Kagoshima
  - Kanazawa University Hospital, Kanazawa
  - Kobe University Hospital, Kobe
  - Kumamoto University Hospital, Kumamoto
  - Kurume University Hospital, Kurume
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Kyoto University Hospital, Kyoto
  - Shinshu University Hospital, Matsumoto
  - Kyorin University Hospital, Mitaka
  - Nagasaki University Hospital, Nagasaki
  - Okayama University Hospital, Okayama
  - National Hospital Organization Okayama Medical Center, Okayama
  - Sapporo Medical University Hospital, Sapporo
  - Hokkaido University Hospital, Sapporo
  - Tohoku University Hospital, Sendai
  - National Cerebral and Cardiovascular Center, Suita-Shi
  - Juntendo University Hospital, Tokyo
  - Mie University Hospital, Tsu
  - University of Tsukuba Hospital, Tsukuba
- Malaysia (2):
  - Institut Jantung Negara (National Heart Institute), Kuala Lumpur
  - Sarawak Heart Center, Kuching
- Mexico (2):
  - Instituto Nacional de Cardiologia Dr. Ignacio Chavez, México
  - Unidad de Investigacion Clinica en Medicina S.C. (UDICEM), Monterrey
- Poland (9):
  - Klinika Kardiologii Z Oddzialem Intensywnego Nadzoru Kardiologicznego UM W Bialymstoku, Bialystok
  - Szpital Uniwersytecki nr 2 im dr Jana Biziela w Bydgoszczy, Klinika Kardiologii, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - GCM SUM I Oddzial Kardiologii, Katowice
  - Oddzial Kardiologii Wojewodzki Szpital Specjalistyczny im W Bieganskiego, Lodz
  - Wojewodzki Szpital Specjalistyczny im. Stefana Kardynala Wyszynskiego SPZOZ, Oddzial Kardiologii, Lublin
  - ECZ Otwock Klinika Kardiologii Klinika Krazenia Plucnego Chorob Zakrzepowo Zatorowych i Kardiologii, Otwock
  - Uniwersytecki Szpital Kliniczny nr 2 PUM Klinika Kardiologii, Szczecin
  - Wojewodzki Szpital Specjalistyczny Oddzial Kardiologiczny, Wroclaw
- Russia (6):
  - Altay Regional Cardiological Dispensary, Barnaul
  - Scientific and Research Institution of Cardiovascular Diseases Complex Problems, Kemerovo
  - National Medical Research Center of Cardiology of MoH of Russian Federation, Moscow
  - GU Moscow Regional Research Clinical Institute n.a. M.F.Vla, Moscva
  - National medical Research Center n.a. V.A.Almazov of MoH of Russian Federation, Saint Petersburg
  - Samara Regional Clinical Cardiological Dispensary, Samara
- South Africa (2):
  - Abdullah, IA, Durban
  - Dr Kalla, Lenasia
- Spain (9):
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Virgen de La Salud, Toledo
  - Hosp. Gral. Univ. Valencia, Valencia
- Taiwan (6):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang-Gung Memorial Hospital, LinKou Branch, Taoyuan District
- Turkey (Türkiye) (12):
  - Cukurova University Medical Faculty, Adana
  - Hacettepe University Medical Faculty, Ankara
  - Ankara University Medical Faculty, Ankara
  - Bursa Yuksek Ihtisas Training and Research Hospital, Bursa
  - Istanbul University - Cerrahpasa Cardiology Institution, Istanbul
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Marmara University Medical Faculty, Istanbul
  - Ege University School of Medicine, Izmir
  - Dokuz Eylul University Hospital, Izmir
  - Kartal Kosuyolu Yuksek Ihtisas Egitim Ve Arastirma Hastanesi, Kartal Istanbul
  - Konya Selcuk University Medical Faculty, Konya
  - Mersin University Medical Faculty, Mersin

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials\transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Fan F, Sun L, Yang Z, Wang L, Wang Q, Li J, Gu H, Xie W, Zhang N, Bin J, Rofael H, Friberg M, Hauser JA. Macitentan Plus Tadalafil Single-Tablet Combination Therapy in Chinese Patients With Pulmonary Arterial Hypertension: A Subgroup Analysis of the A DUE Study. Pulm Circ. 2025 Nov 16;15(4):e70194. doi: 10.1002/pul2.70194. eCollection 2025 Oct. PMID 41250682
- [Derived] Grunig E, Jansa P, Fan F, Hauser JA, Pannaux M, Morganti A, Rofael H, Chin KM. Randomized Trial of Macitentan/Tadalafil Single-Tablet Combination Therapy for Pulmonary Arterial Hypertension. J Am Coll Cardiol. 2024 Jan 30;83(4):473-484. doi: 10.1016/j.jacc.2023.10.045. PMID 38267108
- See also: RRF KOM slides — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=AC-077A301&attachmentIdentifier=6a92fb9d-e152-4929-aa6b-06238109e9a5&fileName=AC-077A301_-_RRF_KOM.pptx&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In open label period, safety was presented using the combination safety set. Combination safety set included all participants randomized to macitentan/tadalafil fixed-dose combination (M/T FDC) in DB period and who received at least 1 dose of M/T FDC in DB treatment and all participants who received at least 1 dose of M/T FDC treatment in OL period.
Groups:
- DB: Treatment-naive and Prior ERA Strata: Macitentan Monotherapy 10 Milligrams (mg): During double-blind (DB) treatment period, participants who were either treatment-naive or on a predefined stable dose of endothelin receptor antagonist (ERA), received one tablet of macitentan 10 mg along with two tablets of placebo matching to tadalafil 20 mg, orally, once daily at Weeks 1 and 2 (titration phase). From Week 3 to 16 (maintenance phase), participants continued to receive one tablet of macitentan 10 mg and two tablets placebo tablet matching to tadalafil 20 mg along with one tablet of placebo matching to macitentan 10 mg and tadalafil 40 mg fixed-dose combination (M/T FDC), orally, once daily.
- DB: Treatment-naive and Prior PDE-5i Strata: Tadalafil Monotherapy 20 mg (2 Tablets*20 mg): During DB treatment period, participants who were either treatment-naive or on a predefined stable dose of phosphodiesterase type-5 inhibitor (PDE-5i), received one tablet (two tablets if already on allowable dose at baseline) of tadalafil 20 mg along with one tablet of placebo matching to macitentan 10 mg and one tablet of placebo matching to tadalafil 20 mg, orally, once daily at Week 1 (titration phase). Participants further received two tablets of tadalafil 20 mg along with one tablet of placebo matching to macitentan 10 mg, orally, once daily at Week 2 (titration phase). From Week 3 to 16 (maintenance phase), participants received two tablets of tadalafil 20 mg along with one tablet of placebo matching to macitentan 10 mg and one tablet of placebo matching to M/T FDC, orally, once daily.
- DB: Treatment-naive and Prior ERA/ PDE-5i Strata: M/T FDC: During DB treatment period, participants who were either treatment-naive or on a predefined stable dose of ERA or PDE-5i, received one tablet of macitentan 10 mg along with one tablet of tadalafil 20 mg and one tablet of placebo matching to tadalafil 20 mg, orally, once daily at Week 1 (uptitration phase). Participants further received one tablet of macitentan 10 mg along with two tablets of tadalafil 20 mg, orally, once daily at Week 2 (uptitration phase). From Week 3 to 16 (maintenance phase), participants received one tablet of placebo matching to macitentan 10 mg along with two tablets of placebo matching to tadalafil 20 mg and one tablet of macitentan 10 mg and tadalafil 40 mg fixed-dose combination (M/T FDC), orally, once daily.
- OL: Treatment-naive and Prior ERA Strata: M/T FDC: After completion of DB phase, participants who were either treatment-naive or on a predefined stable dose of ERA and received macitentan monotherapy during DB phase entered open label (OL) phase. During the OL phase participants received one tablet of macitentan 10 mg along with one tablet of tadalafil 20 mg and one tablet of placebo matching tadalafil 20 mg, orally, once daily for first 7 days (Week 17, titration phase). Subsequently participants received two tablets of tadalafil 20 mg along with one tablet of macitentan 10 mg, orally, once daily for 7 days (Week 18, titration phase). From Weeks 19 to 183 (maintenance phase), participants continued to receive one tablet of M/T FDC, orally, once daily.
- OL: Treatment-naive and Prior PDE-5i Strata: M/T FDC: After completion of DB phase, participants who were either treatment-naive or on a predefined stable dose of PDE-5i and received tadalafil monotherapy during DB phase entered OL phase. During the OL phase participants received one tablet of macitentan 10 mg along with two tablets of tadalafil 20 mg, orally, once daily for the first 2 weeks (Week 17 and Week 18; titration phase). From Weeks 19 to 183 (maintenance phase), participants continued to receive one tablet of M/T FDC, orally, once daily.
- OL: Treatment-naive and Prior ERA/ PDE-5i Strata: M/T FDC: After completion of DB phase, participants who were either treatment-naive or on a predefined stable dose of ERA or PDE-5i and received M/T FDC during DB phase entered OL phase. During the OL phase participants received one tablet macitentan 10 mg along with two tablets of tadalafil 20 mg, orally, once daily for 2 weeks (Week 17 and Week 18; titration phase). From Weeks 19 to 183 (maintenance phase), participants continued to receive one tablet of M/T FDC, orally, once daily.
Period: DB Treatment Period (Week 1 to Week 16)
Arm/Group | DB: Treatment-naive and Prior ERA Strata: Macitentan Monotherapy 10 Milligrams (mg) | DB: Treatment-naive and Prior PDE-5i Strata: Tadalafil Monotherapy 20 mg (2 Tablets*20 mg) | DB: Treatment-naive and Prior ERA/ PDE-5i Strata: M/T FDC | OL: Treatment-naive and Prior ERA Strata: M/T FDC | OL: Treatment-naive and Prior PDE-5i Strata: M/T FDC | OL: Treatment-naive and Prior ERA/ PDE-5i Strata: M/T FDC
Started | 35 | 44 | 108 (Treatment naive participants are counted once as enrolled but contributed to data twice based on strata (prior ERA/PDE-5i strata). 108 includes one participant who did not receive treatment.) | 0 | 0 | 0
Treated (Safety Analysis Set) | 35 | 44 | 107 | 0 | 0 | 0
Treatment Naive and Prior ERA Strata: M/T FDC | 0 | 0 | 71 | 0 | 0 | 0
Treatment Naive and Prior PDE-5i Strata: M/T FDC | 0 | 0 | 87 | 0 | 0 | 0
Completed | 35 | 43 | 99 | 0 | 0 | 0
Not Completed | 0 | 1 | 9 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 3 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 4 | 0 | 0 | 0
Period: OL Treatment Period (Week 17 to Week189)
Arm/Group | DB: Treatment-naive and Prior ERA Strata: Macitentan Monotherapy 10 Milligrams (mg) | DB: Treatment-naive and Prior PDE-5i Strata: Tadalafil Monotherapy 20 mg (2 Tablets*20 mg) | DB: Treatment-naive and Prior ERA/ PDE-5i Strata: M/T FDC | OL: Treatment-naive and Prior ERA Strata: M/T FDC | OL: Treatment-naive and Prior PDE-5i Strata: M/T FDC | OL: Treatment-naive and Prior ERA/ PDE-5i Strata: M/T FDC
Started | 0 | 0 | 0 | 35 | 43 | 91
Completed | 0 | 0 | 0 | 30 | 38 | 76
Not Completed | 0 | 0 | 0 | 5 | 5 | 15
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 4 | 7
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Initiated prohibited medication | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Non-compliance with study drug | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Technical problems | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Family problems | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set (SAS) included all randomized participants who received at least one dose of study treatment (for participants on FDC, at least one dose of either macitentan or tadalafil).
Groups:
- Total: Total of all reporting groups
Arm/Group | DB: Treatment-naive and Prior ERA Strata: Macitentan Monotherapy 10 Milligrams (mg) | DB: Treatment-naive and Prior PDE-5i Strata: Tadalafil Monotherapy 20 mg (2 Tablets*20 mg) | DB: Treatment-naive and Prior ERA/ PDE-5i Strata: M/T FDC | Total
Number analyzed (Participants) | 35 | 44 | 107 | 186
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 34 | 87 | 148
  >=65 years | 8 | 10 | 20 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (15.85) | 53.1 (13.66) | 48.7 (15.78) | 50.2 (15.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 34 | 82 | 145
  Male | 6 | 10 | 25 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 8 | 15
  Not Hispanic or Latino | 30 | 39 | 95 | 164
  Unknown or Not Reported | 3 | 0 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 12 | 11 | 36 | 59
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 2 | 5
  White | 20 | 29 | 66 | 115
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 2 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  BRAZIL | 5 | 3 | 4 | 12
  BULGARIA | 0 | 2 | 2 | 4
  CANADA | 0 | 1 | 1 | 2
  CHINA | 5 | 5 | 13 | 23
  GERMANY | 2 | 4 | 7 | 13
  ITALY | 1 | 1 | 4 | 6
  JAPAN | 1 | 1 | 6 | 8
  MALAYSIA | 1 | 2 | 10 | 13
  MEXICO | 2 | 2 | 6 | 10
  POLAND | 3 | 2 | 7 | 12
  RUSSIAN FEDERATION | 1 | 0 | 10 | 11
  SOUTH AFRICA | 3 | 2 | 1 | 6
  SPAIN | 3 | 2 | 3 | 8
  TAIWAN | 3 | 2 | 6 | 11
  TURKEY | 1 | 2 | 14 | 17
  UNITED STATES | 4 | 13 | 13 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Pulmonary Vascular Resistance (PVR) Expressed as the Ratio of Geometric Means of End of Double-blind Treatment (EDBT) to Baseline
Description: Change in PVR expressed as the ratio of geometric means of EDBT to baseline were reported.
Time Frame: Baseline, EDBT (up to 16 weeks)
Population: The full analysis set (FAS) included all randomized participants who received at least one dose of study treatment (for participants on FDC, at least one dose of either macitentan or tadalafil). Treatment-naive participants randomized to both M/T FDC arms (ERA and PDE-5i strata) are counted twice as per planned analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Groups:
- DB: Treatment-naive And Prior ERA Strata: Macitentan Monotherapy 10 Milligrams (mg): During double-blind (BD) treatment period, participants who were either treatment-naive or on a predefined stable dose of endothelin receptor antagonist (ERA), received one tablet of macitentan 10 mg along with two tablets of placebo matching to tadalafil 20 mg, orally, once daily at Weeks 1 and 2 (titration phase). From Week 3 to 16 (maintenance phase), participants continued to receive one tablet of macitentan 10 mg and two tablets placebo tablet matching to tadalafil 20 mg along with one tablet of placebo matching to macitentan 10 mg and tadalafil 40 mg fixed-dose combination (M/T FDC), orally, once daily.
- DB: Treatment-naive And Prior ERA Strata: M/T FDC: During DB treatment period, participants who were either treatment-naive or on a predefined stable dose of ERA, received one tablet of macitentan 10 mg along with one tablet of tadalafil 20 mg and one tablet of placebo matching to tadalafil 20 mg, orally, once daily at Week 1 (uptitration phase). Participants further received one tablet of macitentan 10 mg along with two tablets of tadalafil 20 mg, orally, once daily at Week 2 (uptitration phase). From Week 3 to 16 (maintenance phase), participants received one tablet of placebo matching to macitentan 10 mg along with two tablets of placebo matching to tadalafil 20 mg and one tablet of macitentan 10 mg and tadalafil 40 mg fixed-dose combination (M/T FDC), orally, once daily.
- DB: Treatment-naive And Prior PDE-5i Strata: M/T FDC: During DB treatment period, participants who were either treatment-naive or on a predefined stable dose of PDE-5i, received one tablet of macitentan 10 mg along with one tablet of tadalafil 20 mg and one tablet of placebo matching to tadalafil 20 mg, orally, once daily at Week 1 (uptitration phase). Participants further received one tablet of macitentan 10 mg along with two tablets of tadalafil 20 mg, orally, once daily at Week 2 (uptitration phase). From Week 3 to 16 (maintenance phase), participants received one tablet of placebo matching to macitentan 10 mg along with two tablets of placebo matching to tadalafil 20 mg and one tablet of macitentan 10 mg and tadalafil 40 mg fixed-dose combination (M/T FDC), orally, once daily.
Arm/Group | DB: Treatment-naive And Prior ERA Strata: Macitentan Monotherapy 10 Milligrams (mg) | DB: Treatment-naive And Prior ERA Strata: M/T FDC | DB: Treatment-naive And Prior PDE-5i Strata: Tadalafil Monotherapy 20 mg (2 Tablets*20 mg) | DB: Treatment-naive And Prior PDE-5i Strata: M/T FDC
Number analyzed (Participants) | 35 | 70 | 44 | 86
Ratio | 0.77 [0.69 to 0.87] | 0.55 [0.50 to 0.60] | 0.78 [0.72 to 0.84] | 0.56 [0.52 to 0.60]
Statistical Analysis 1: Comparison: DB: Treatment-naive And Prior ERA Strata: Macitentan Monotherapy 10 Milligrams (mg) vs DB: Treatment-naive And Prior ERA Strata: M/T FDC; Test type: Superiority; p < 0.0001, ANCOVA; Geometric Mean Ratio = 0.71, 95% CI 2-sided [0.61 to 0.82]
Statistical Analysis 2: Comparison: DB: Treatment-naive And Prior PDE-5i Strata: Tadalafil Monotherapy 20 mg (2 Tablets*20 mg) vs DB: Treatment-naive And Prior PDE-5i Strata: M/T FDC; Test type: Superiority; p < 0.0001, ANCOVA; Geometric Mean Ratio = 0.72, 95% CI 2-sided [0.64 to 0.80]

2. Secondary Outcome: Change From Baseline to EDBT in 6-minutes Walking Distance (6MWD)
Description: Change from baseline to EDBT in 6MWD were reported. 6MWD was measured by 6-minute walk test (6MWT). The test measured the distance an individual was able to walk over a total of six minutes on a hard, flat surface with no obstacles. The goal was for the individual to walk as far as possible in 6 minutes.
Time Frame: Baseline, EDBT (Week 16)
Population: The FAS included all randomized participants who received at least one dose of study treatment (for participants on FDC, at least one dose of either macitentan or tadalafil). Treatment-naive participants randomized to both macitentan 10 mg and tadalafil 40 mg fixed-dose combination (M/T FDC) arms (ERA and PDE-5i strata) are counted twice as per planned analysis.
Measure: Mean (Standard Deviation); unit: Meters
Groups:
- DB: Treatment-naive And Prior ERA Strata: Macitentan 10 Milligrams (mg): During double-blind treatment period, participants who were either treatment-naive or on a predefined stable dose of endothelin receptor antagonist (ERA), received one tablet of macitentan 10 mg along with two tablets of placebo matching to tadalafil 20 mg, orally, once daily at Weeks 1 and 2 (titration phase). From Week 3 to 16 (maintenance phase), participants continued to receive one tablet of macitentan 10 mg and two tablets placebo tablet matching to tadalafil 20 mg along with one tablet of placebo matching to macitentan 10 mg and tadalafil 40 mg fixed-dose combination (M/T FDC), orally, once daily.
- DB: Treatment-naive And Prior PDE-5i Strata: M/T FDC: During double-blind treatment period, participants who were either treatment-naive or on a predefined stable dose of PDE-5i, received one tablet of macitentan 10 mg along with one tablet of tadalafil 20 mg and one tablet of placebo matching to tadalafil 20 mg, orally, once daily at Week 1 (uptitration phase). Participants further received one tablet of macitentan 10 mg along with two tablets of tadalafil 20 mg, orally, once daily at Week 2 (uptitration phase). From Week 3 to 16 (maintenance phase), participants received one tablet of placebo matching to macitentan 10 mg along with two tablets of placebo matching to tadalafil 20 mg and one tablet of macitentan 10 mg and tadalafil 40 mg fixed-dose combination (M/T FDC), orally, once daily.
Arm/Group | DB: Treatment-naive And Prior ERA Strata: Macitentan 10 Milligrams (mg) | DB: Treatment-naive And Prior ERA Strata: M/T FDC | DB: Treatment-naive And Prior PDE-5i Strata: Tadalafil Monotherapy 20 mg (2 Tablets*20 mg) | DB: Treatment-naive And Prior PDE-5i Strata: M/T FDC
Number analyzed (Participants) | 35 | 70 | 44 | 86
Meters | 38.5 (70.42) | 52.9 (88.23) | 15.9 (45.04) | 43.4 (78.03)
Statistical Analysis 1: Comparison: DB: Treatment-naive And Prior ERA Strata: Macitentan 10 Milligrams (mg) vs DB: Treatment-naive And Prior ERA Strata: M/T FDC; Test type: Superiority; p = 0.3802, ANCOVA; Geometric Mean Ratio = 16.04, 95% CI 2-sided [-17.0 to 49.08]
Statistical Analysis 2: Comparison: DB: Treatment-naive And Prior PDE-5i Strata: Tadalafil Monotherapy 20 mg (2 Tablets*20 mg) vs DB: Treatment-naive And Prior PDE-5i Strata: M/T FDC; Test type: Superiority; p = 0.0591, ANCOVA; Geometric Mean Ratio = 25.37, 95% CI 2-sided [-0.93 to 51.59]

3. Secondary Outcome: Change From Baseline in Pulmonary Arterial Hypertension Symptoms and Impact (PAH-SYMPACT) in Cardiopulmonary Symptom Domain Scores to EDBT
Description: Change from baseline in PAH-SYMPACT in cardiopulmonary symptom domain scores to EDBT were reported. PAH-SYMPACT was a pulmonary arterial hypertension (PAH)-specific patient-reported outcomes questionnaire that consists of 11 symptoms items, 11 impacts items and 1 item on oxygen use. The symptom items were divided into cardiopulmonary and cardiovascular domains, and the impact items were divided into physical and emotional/cognitive domains. Cardiopulmonary symptoms contain 6 items; shortness of breath, fatigue, lack of energy, swelling in ankles or legs, swelling in stomach area, and cough. Scores for the individual items were reported on a 5-point Likert scale, ranging from 0 (no symptom at all) to 4 (very severe symptoms), with higher scores indicated greater symptom severity.
Time Frame: Baseline, EDBT (Week 16)
Population: The PAH-SYMPACT symptoms analysis set included all participants included in the FAS for whom at least one baseline value of symptoms domain was provided. Treatment-naive participants randomized to both M/T FDC arms (ERA and PDE-5i strata) were counted twice as per planned analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | DB: Treatment-naive And Prior ERA Strata: Macitentan 10 Milligrams (mg) | DB: Treatment-naive And Prior ERA Strata: M/T FDC | DB: Treatment-naive And Prior PDE-5i Strata: Tadalafil Monotherapy 20 mg (2 Tablets*20 mg) | DB: Treatment-naive And Prior PDE-5i Strata: M/T FDC
Number analyzed (Participants) | 33 | 66 | 42 | 81
Score on a scale | -0.14 (0.478) | -0.20 (0.394) | -0.13 (0.554) | -0.15 (0.404)

4. Secondary Outcome: Change From Baseline in Pulmonary Arterial Hypertension Symptoms and Impact (PAH-SYMPACT) in Cardiovascular Symptom Domain Scores to EDBT
Description: Change from baseline in PAH-SYMPACT in cardiovascular symptom domain scores to EDBT were reported. PAH-SYMPACT is a PAH-specific patient-reported outcomes questionnaire that consists of 11 symptoms items, 11 impacts items and 1 item on oxygen use. The symptom items were divided into cardiopulmonary and cardiovascular domains, and the impact items were divided into physical and emotional/cognitive domains. Cardiovascular symptoms contain 5 items; heart palpitations (heart fluttering), rapid heartbeat, chest pain, chest tightness, and lightheadedness. Scores for the individual items were reported on a 5-point Likert scale, ranging from 0 (no symptom at all) to 4 (very severe symptom), with higher scores indicated greater symptom severity.
Time Frame: Baseline, EDBT (Week 16)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | DB: Treatment-naive And Prior ERA Strata: Macitentan 10 Milligrams (mg) | DB: Treatment-naive And Prior ERA Strata: M/T FDC | DB: Treatment-naive And Prior PDE-5i Strata: Tadalafil Monotherapy 20 mg (2 Tablets*20 mg) | DB: Treatment-naive And Prior PDE-5i Strata: M/T FDC
Number analyzed (Participants) | 33 | 66 | 42 | 81
Score on a scale | -0.14 (0.473) | -0.15 (0.349) | -0.18 (0.612) | -0.10 (0.318)

5. Secondary Outcome: Percentage of Participants With Absence of Worsening in World Health Organization (WHO) Functional Class (FC) From Baseline at EDBT
Description: Percentage of participants with absence of worsening in FC from baseline to EDBT were reported. The study was adaptive with two stages: Stage 1 and Stage 2. WHO functional classification (FC), PAH range from Class I (no limitation in physical activity, no dyspnea or fatigue, chest pain, or near syncope with normal activity), Class II (slight limitation of physical activity), Class III (marked limitation of physical activity), Class IV (cannot perform a physical activity without any symptoms, dyspnea and/or fatigue at rest).
Time Frame: At Week 16 (EDBT)
Population: The FAS included all randomized participants who received at least one dose of study treatment (for participants on FDC, at least one dose of either macitentan or tadalafil). Treatment-naive participants randomized to both M/T FDC arms (ERA and PDE-5i strata) are counted twice as per planned analysis. Here, 'N' overall (number of participants analyzed) signifies the number of participants evaluable, "n" (number analyzed) =number of participants evaluable for specified category.
Measure: Number; unit: Percentage of participants
Arm/Group | DB: Treatment-naive And Prior ERA Strata: Macitentan 10 Milligrams (mg) | DB: Treatment-naive And Prior ERA Strata: M/T FDC | DB: Treatment-naive And Prior PDE-5i Strata: Tadalafil Monotherapy 20 mg (2 Tablets*20 mg) | DB: Treatment-naive And Prior PDE-5i Strata: M/T FDC
Number analyzed (Participants) | 18 | 38 | 22 | 47
Percentage of participants
  Stage: 1 : Class I | 5.6 [lower limit 0.590] | 5.3 [lower limit 0.561] | 4.5 [lower limit 0.522] | 12.8 [lower limit 0.546]
  Stage: 1 : Class II | 55.6 | 57.9 | 63.6 | 59.6
  Stage: 1 : Class III | 38.9 | 23.7 | 31.8 | 25.5
  Stage: 1 : Class IV | 0 | 0 | 0 | 0
  Stage: 1 : Missing | 0 | 13.2 | 0 | 2.1
  Stage: 2 : Class I: number analyzed (Participants) | 17 | 32 | 22 | 39
  Stage: 2 : Class I | 11.8 | 9.4 | 9.1 | 7.7
  Stage: 2 : Class II: number analyzed (Participants) | 17 | 32 | 22 | 39
  Stage: 2 : Class II | 52.9 | 75.0 | 54.5 | 61.5
  Stage: 2: Class III: number analyzed (Participants) | 17 | 32 | 22 | 39
  Stage: 2: Class III | 35.3 | 15.6 | 36.4 | 25.6
  Stage: 2 : Class IV: number analyzed (Participants) | 17 | 32 | 22 | 39
  Stage: 2 : Class IV | 0 | 0 | 0 | 0
  Stage: 2 : Missing: number analyzed (Participants) | 17 | 32 | 22 | 39
  Stage: 2 : Missing | 0 | 0 | 0 | 5.1

ADVERSE EVENTS:
Time Frame: DB: All-cause mortality: From baseline (pre-dose Day 1) to Week 16; SAE and other AEs: From Day 1 to Week 16; OL phase: From Week 16 up to 35 days after last dose (Week 189)
Description: All-cause mortality: all randomized. SAE/Other AEs: DB: all treated participants. OL: combined safety set was used. Treatment naive participants in both M/T FDC arms (ERA/PDE-5i strata) counted twice per planned analysis. Per plan, for participants treated with M/T FDC in DB, combined data from DB and OL phase collected and analyzed in OL. During OL phase, objective was to analyze safety for M/T FDC irrespective of strata, hence data for combined strata is reported in DB + OL arm, per plan.
Groups:
- DB + OL: Treatment-naive and Prior ERA/ PDE-5i Strata: M/T FDC: During DB treatment period, participants who were either treatment-naive or on a predefined stable dose of ERA or PDE-5i, received macitentan 10 mg along with tadalafil 20 mg and placebo matching to tadalafil 20 mg, orally, once daily at Week 1 (uptitration phase). Participants further received one tablet of macitentan 10 mg along with two tablets of tadalafil 20 mg, orally, once daily at Week 2 (uptitration phase). From Week 3 to 16 (maintenance phase), participants received one tablet of placebo matching to macitentan 10 mg along with two tablets of placebo matching to tadalafil 20 mg and one tablet of macitentan 10 mg and tadalafil 40 mg fixed-dose combination (M/T FDC), orally, once daily. After completion of DB phase, participants who were either treatment-naive or on a predefined stable dose of ERA or PDE-5i and received M/T FDC during DB phase entered OL phase. During the OL phase participants received one tablet macitentan 10 mg along with two tablets of tadalafil 20 mg, orally, once daily for 2 weeks (Week 17 and Week 18; titration phase). From Weeks 19 to 183 (maintenance phase), participants continued to receive one tablet of M/T FDC, orally, once daily.
Arm/Group | DB: Treatment-naive and Prior ERA Strata: Macitentan Monotherapy 10 Milligrams (mg) | DB: Treatment-naive And Prior ERA Strata: M/T FDC | DB: Treatment-naive And Prior PDE-5i Strata: Tadalafil Monotherapy 20 mg (2 Tablets*20 mg) | DB: Treatment-naive And Prior PDE-5i Strata: M/T FDC | DB: Treatment-naive and Prior ERA/ PDE-5i Strata: M/T FDC | OL: Treatment-naive and Prior ERA Strata: M/T FDC | OL: Treatment-naive and Prior PDE-5i Strata: M/T FDC | DB + OL: Treatment-naive and Prior ERA/ PDE-5i Strata: M/T FDC
All-Cause Mortality (participants affected / at risk) | 0/35 | 2/71 | 0/44 | 2/87 | 3/108 | 0/35 | 2/43 | 9/107
Serious Adverse Events (participants affected / at risk) | 3/35 | 11/70 | 4/44 | 12/86 | 15/107 | 10/35 | 13/43 | 39/107
Other Adverse Events (participants affected / at risk) | 16/35 | 49/70 | 31/44 | 58/86 | 72/107 | 28/35 | 38/43 | 89/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB: Treatment-naive and Prior ERA Strata: Macitentan Monotherapy 10 Milligrams (mg) (N=35) | DB: Treatment-naive And Prior ERA Strata: M/T FDC (N=70) | DB: Treatment-naive And Prior PDE-5i Strata: Tadalafil Monotherapy 20 mg (2 Tablets*20 mg) (N=44) | DB: Treatment-naive And Prior PDE-5i Strata: M/T FDC (N=86) | DB: Treatment-naive and Prior ERA/ PDE-5i Strata: M/T FDC (N=107) | OL: Treatment-naive and Prior ERA Strata: M/T FDC (N=35) | OL: Treatment-naive and Prior PDE-5i Strata: M/T FDC (N=43) | DB + OL: Treatment-naive and Prior ERA/ PDE-5i Strata: M/T FDC (N=107)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1
Normochromic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angina Pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial Flutter (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Cardiac Failure (Cardiac disorders) | 0 | 2 | 1 | 1 | 2 | 0 | 0 | 2
Cor Pulmonale (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1
Left Ventricular Failure (Cardiac disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Right Ventricular Failure (Cardiac disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 4
Sinus Node Dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retinal Vein Occlusion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colitis Ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hiatus Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Large Intestine Polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophageal Ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tongue Cyst (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Varices Oesophageal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest Pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral Swelling (General disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1
Swelling Face (General disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1
Hepatic Cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Portal Hypertension (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abscess Bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Covid-19 (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 5
Covid-19 Pneumonia (Infections and infestations) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 2
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis Clostridial (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Parainfluenzae Virus Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 3
Pneumonia Viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rhinovirus Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Staphylococcal Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Jaw Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Patella Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Greater Trochanteric Pain Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Systemic Scleroderma (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mucinous Cystadenocarcinoma Ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Cerebral Infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Horner's Syndrome (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Glomerulonephritis Membranous (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal Impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Endometrial Hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Intermenstrual Bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ovarian Cyst Ruptured (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Uterine Polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Autoimmune Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 2 | 0 | 0 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary Arterial Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Pulmonary Veno-Occlusive Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB: Treatment-naive and Prior ERA Strata: Macitentan Monotherapy 10 Milligrams (mg) (N=35) | DB: Treatment-naive And Prior ERA Strata: M/T FDC (N=70) | DB: Treatment-naive And Prior PDE-5i Strata: Tadalafil Monotherapy 20 mg (2 Tablets*20 mg) (N=44) | DB: Treatment-naive And Prior PDE-5i Strata: M/T FDC (N=86) | DB: Treatment-naive and Prior ERA/ PDE-5i Strata: M/T FDC (N=107) | OL: Treatment-naive and Prior ERA Strata: M/T FDC (N=35) | OL: Treatment-naive and Prior PDE-5i Strata: M/T FDC (N=43) | DB + OL: Treatment-naive and Prior ERA/ PDE-5i Strata: M/T FDC (N=107)
Anaemia (Blood and lymphatic system disorders) | 0 | 6 | 0 | 6 | 8 | 4 | 5 | 13
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 2 | 2 | 0 | 2 | 6
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2
Palpitations (Cardiac disorders) | 1 | 1 | 2 | 2 | 3 | 1 | 3 | 7
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 6 | 5 | 5 | 0 | 2 | 7
Dyspepsia (Gastrointestinal disorders) | 0 | 4 | 3 | 4 | 4 | 0 | 1 | 4
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2 | 3 | 0 | 4
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1 | 3 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 3
Nausea (Gastrointestinal disorders) | 0 | 5 | 3 | 4 | 6 | 1 | 1 | 8
Vomiting (Gastrointestinal disorders) | 0 | 3 | 2 | 4 | 4 | 0 | 2 | 9
Fatigue (General disorders) | 1 | 2 | 1 | 2 | 3 | 0 | 0 | 7
Non-Cardiac Chest Pain (General disorders) | 0 | 2 | 3 | 2 | 3 | 0 | 1 | 3
Oedema Peripheral (General disorders) | 4 | 9 | 5 | 12 | 14 | 1 | 5 | 16
Peripheral Swelling (General disorders) | 1 | 6 | 0 | 6 | 6 | 1 | 0 | 7
Pyrexia (General disorders) | 0 | 2 | 0 | 4 | 4 | 0 | 5 | 7
Covid-19 (Infections and infestations) | 2 | 1 | 2 | 2 | 2 | 7 | 10 | 25
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 3 | 3 | 2 | 2 | 7
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 2
Suspected Covid-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 2 | 0 | 1 | 2 | 5 | 6 | 5
Urinary Tract Infection (Infections and infestations) | 0 | 2 | 0 | 0 | 2 | 2 | 4 | 6
Blood Glucose Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Haemoglobin Decreased (Investigations) | 0 | 3 | 0 | 8 | 8 | 4 | 1 | 13
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 4 | 1 | 4 | 4 | 0 | 0 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 2 | 3 | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4 | 4 | 4 | 3 | 3 | 8
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 5 | 4 | 3 | 5 | 2 | 2 | 7
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 5 | 2 | 4 | 6 | 5 | 2 | 7
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 4 | 2 | 3 | 1 | 1 | 6
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 1 | 3 | 3 | 2 | 1 | 6
Headache (Nervous system disorders) | 6 | 12 | 6 | 14 | 18 | 3 | 2 | 23
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 2 | 6 | 6 | 2 | 5 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 2 | 2 | 0 | 7 | 5
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 3 | 4 | 1 | 2 | 6
Flushing (Vascular disorders) | 2 | 3 | 0 | 3 | 3 | 0 | 0 | 4
Hypotension (Vascular disorders) | 0 | 5 | 0 | 4 | 7 | 1 | 1 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related publication written independently by investigators must be submitted to the sponsor for review at least 30 days prior to submission for publication or presentation at a congress. Upon review, the sponsor may provide comments, and may also request alterations and/or deletions for the sole purpose of protecting its confidential information and/or patent rights. Neither the institution nor the investigator should permit publication during such a review period.

DOCUMENTS (2):
  • Study Protocol (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/93/NCT03904693/Prot_002.pdf
  • Statistical Analysis Plan (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/93/NCT03904693/SAP_003.pdf